CLINICAL TRIAL: NCT03927898
Title: Phase II Study of Toripalimab (JS001) Plus Stereotactic Body Radiotherapy in Colorectal Cancer Patients With Oligometastasis
Brief Title: Phase II Study of Toripalimab Plus Stereotactic Body Radiotherapy in Colorectal Cancer Patients With Oligometastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., Professor of Dept.of Radiation Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-223/1781
Record Dates: First submitted 2019-04-09; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — toripalimab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: All enrolled patients will receive Toripalimab following stereotactic body radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+Toripalimab (Experimental): Participants received SBRT (BED>80Gy) to oligometastatic lesions and then receive Toripalimab (240mg)/q3w till progression of disease.
  Interventions: Drug: Toripalimab; Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Drug: Toripalimab — Participants receive Toripalimab (240mg)/q3w till progression of disease after SBRT
Radiation: Stereotactic Body Radiotherapy — Participants receive SBRT (BED>80Gy) to oligometastatic lesions followed by Toripalimab (240mg)/q3w

SUMMARY:
Metastatic colorectal cancer is one of the common malignant tumors and the overall prognosis is poor. The introduction of immune-checkpoint inhibition (ICI) has led to a paradigm shift in the treatment of patients with metastatic cancer. Stereotactic body radiation therapy (SBRT) delivers a large dose of radiation to the tumor target with high precision while sparing irradiation of the surrounding normal tissues. It is suggested that SBRT could be the most appropriate radiotherapy modality to be combined with immunotherapy since it induces the expression of a series of cytokines and new tumour-associated antigens (TAAs) and is more likely to cause intense immune response and exert an abscopal effect than conventional radiotherapy.

Thus, this study is to explore the use of SBRT in combination with ICI in colorectal cancer patients with oligometastasis, in order to get better local and systemic tumor control and improve progress-free survival (PFS).

DETAILED DESCRIPTION:
The investigators plan to recruit patients with mCRC, who have received first-line systemic therapy for more than 3 months and achieved PR/SD. Than all the patients will receive SBRT followed by ICI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18-75 years old , Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
2. Histologically confirmed CRC , metastatic CRC , subjects have received first-line systemic therapy for more than 3 months and achieved PR/SD, the interval between last systemic therapy and SBRT is≥4 weeks
3. The primary site has been controlled by surgery
4. Patient has at least 1 lesion of measurable metastatic disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and iRECIST , and who can achieve the status of non evidence of disease after local ablative therapy. The number of lesion is ≤ 5, the maximum diameter of the lesion is ≤5cm ,
5. All metastatic lesions are amenable to SBRT with BED≥80Gy in 3 to 5 fractions;
6. Have a life expectancy of at least 6 months
7. Adequate organ function, as defined by the following:

   Hemoglobin ≥ 100 g/L; White blood cell count (WBC) ≥3.5×109/L , Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelets ≥75×109/L; Serum creatinine ≤ 1.0 x institutional upper limit of normal (ULN) ; Blood Urea Nitrogen(BUN) ≤ 1.0 x institutional (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 x institutional ULN ALkaline Phosphatase (ALP) ≤ 1.5 x institutional ULN Serum total bilirubin (TBIL) ≤1.5 x institutional ULN Urine protein is negative , Coagulation function is normal
8. patients and his/her mate must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug；
9. Patient must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Serious autoimmune disease at the discretion of the treating attending，subjects with leukodermia，allergic asthma syndrome will not be excluded from the study.
2. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Has evidence of interstitial lung disease or active, non-infectious pneumonitis requiring systemic steroids.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study Day 1 of the trial treatment.
5. Has a known additional malignancy，subjects with basal cell carcinoma (BCC)， squamous cell carcinoma of skin and carcinoma in situ of cervix will not be excluded from the study.
6. Has received a vaccine within 30 days prior to study Day 1 of the trial treatment or will receive a vaccine after the trial treatment; active HBV，HCV infection
7. Has received systemic therapy within 4 weeks prior to study Day 1 of the trial treatment or who has not recovered from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy or myelosuppression are an exception to this criterion and may qualify for the study.
8. Any underlying medical or psychiatric condition: partial endocrine organ deficiencies , serious cardiac，pulmonary，renal disease，active infectious disease.
9. Active diverticulitis, intra-abdominal abscess, Gastrointestinal (GI) obstruction, abdominal carcinomatosis , frequent diarrhea or other known risk factors for bowel perforation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
1 year Progression-Free-Survival (PFS) | 1 year
  1 year PFS

SECONDARY OUTCOMES:
Grade 3-5 acute adverse events | 6 months since last treatment of Toripalimab
  Grade 3-5 acute adverse events
Objective response rate | At the end of 4 cycles of Toripalimab (each cycle is 21 days)
  Objective response rate
2 year local control rate | 2 year
  2 year local control rate
2 year overall survival | 2 year
  2 year overall survival
T cell receptor repertoire and T cell clones in peripheral blood | At the end of 6 cycles of Toripalimab (each cycle is 21 days)
  Change of T cell receptor repertoire and T cell clones in peripheral blood
Expression of PD-1, ki-67 on T cell | At the end of 6 cycles of Toripalimab (each cycle is 21 days)
  Change of expression of PD-1, ki-67 on T cell
Expression of PD-L1 on Exosomes in peripheral blood | At the end of 6 cycles of Toripalimab (each cycle is 21 days)
  Change of expression of PD-L1 on Exosomes in peripheral blood
Expression of PD-L1 on circulation tumor cell | At the end of 6 cycles of Toripalimab (each cycle is 21 days)
  Change of expression of PD-L1 on circulation tumor cell

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Background] Petrelli F, Comito T, Barni S, Pancera G, Scorsetti M, Ghidini A; SBRT for CRC liver metastases. Stereotactic body radiotherapy for colorectal cancer liver metastases: A systematic review. Radiother Oncol. 2018 Dec;129(3):427-434. doi: 10.1016/j.radonc.2018.06.035. Epub 2018 Jul 9. PMID 29997034
- [Background] Joo JH, Park JH, Kim JC, Yu CS, Lim SB, Park IJ, Kim TW, Hong YS, Kim KP, Yoon SM, Park J, Kim JH. Local Control Outcomes Using Stereotactic Body Radiation Therapy for Liver Metastases From Colorectal Cancer. Int J Radiat Oncol Biol Phys. 2017 Nov 15;99(4):876-883. doi: 10.1016/j.ijrobp.2017.07.030. Epub 2017 Jul 31. PMID 29063852
- [Background] Luke JJ, Lemons JM, Karrison TG, Pitroda SP, Melotek JM, Zha Y, Al-Hallaq HA, Arina A, Khodarev NN, Janisch L, Chang P, Patel JD, Fleming GF, Moroney J, Sharma MR, White JR, Ratain MJ, Gajewski TF, Weichselbaum RR, Chmura SJ. Safety and Clinical Activity of Pembrolizumab and Multisite Stereotactic Body Radiotherapy in Patients With Advanced Solid Tumors. J Clin Oncol. 2018 Jun 1;36(16):1611-1618. doi: 10.1200/JCO.2017.76.2229. Epub 2018 Feb 13. PMID 29437535
- [Background] Lee Y, Auh SL, Wang Y, Burnette B, Wang Y, Meng Y, Beckett M, Sharma R, Chin R, Tu T, Weichselbaum RR, Fu YX. Therapeutic effects of ablative radiation on local tumor require CD8+ T cells: changing strategies for cancer treatment. Blood. 2009 Jul 16;114(3):589-95. doi: 10.1182/blood-2009-02-206870. Epub 2009 Apr 6. PMID 19349616
- [Background] Tang C, Welsh JW, de Groot P, Massarelli E, Chang JY, Hess KR, Basu S, Curran MA, Cabanillas ME, Subbiah V, Fu S, Tsimberidou AM, Karp D, Gomez DR, Diab A, Komaki R, Heymach JV, Sharma P, Naing A, Hong DS. Ipilimumab with Stereotactic Ablative Radiation Therapy: Phase I Results and Immunologic Correlates from Peripheral T Cells. Clin Cancer Res. 2017 Mar 15;23(6):1388-1396. doi: 10.1158/1078-0432.CCR-16-1432. Epub 2016 Sep 20. PMID 27649551
- [Background] Kwon ED, Drake CG, Scher HI, Fizazi K, Bossi A, van den Eertwegh AJ, Krainer M, Houede N, Santos R, Mahammedi H, Ng S, Maio M, Franke FA, Sundar S, Agarwal N, Bergman AM, Ciuleanu TE, Korbenfeld E, Sengelov L, Hansen S, Logothetis C, Beer TM, McHenry MB, Gagnier P, Liu D, Gerritsen WR; CA184-043 Investigators. Ipilimumab versus placebo after radiotherapy in patients with metastatic castration-resistant prostate cancer that had progressed after docetaxel chemotherapy (CA184-043): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2014 Jun;15(7):700-12. doi: 10.1016/S1470-2045(14)70189-5. Epub 2014 May 13. PMID 24831977
- [Background] Huang AC, Postow MA, Orlowski RJ, Mick R, Bengsch B, Manne S, Xu W, Harmon S, Giles JR, Wenz B, Adamow M, Kuk D, Panageas KS, Carrera C, Wong P, Quagliarello F, Wubbenhorst B, D'Andrea K, Pauken KE, Herati RS, Staupe RP, Schenkel JM, McGettigan S, Kothari S, George SM, Vonderheide RH, Amaravadi RK, Karakousis GC, Schuchter LM, Xu X, Nathanson KL, Wolchok JD, Gangadhar TC, Wherry EJ. T-cell invigoration to tumour burden ratio associated with anti-PD-1 response. Nature. 2017 May 4;545(7652):60-65. doi: 10.1038/nature22079. Epub 2017 Apr 10. PMID 28397821
- [Background] Chen G, Huang AC, Zhang W, Zhang G, Wu M, Xu W, Yu Z, Yang J, Wang B, Sun H, Xia H, Man Q, Zhong W, Antelo LF, Wu B, Xiong X, Liu X, Guan L, Li T, Liu S, Yang R, Lu Y, Dong L, McGettigan S, Somasundaram R, Radhakrishnan R, Mills G, Lu Y, Kim J, Chen YH, Dong H, Zhao Y, Karakousis GC, Mitchell TC, Schuchter LM, Herlyn M, Wherry EJ, Xu X, Guo W. Exosomal PD-L1 contributes to immunosuppression and is associated with anti-PD-1 response. Nature. 2018 Aug;560(7718):382-386. doi: 10.1038/s41586-018-0392-8. Epub 2018 Aug 8. PMID 30089911
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Hanna GG, Murray L, Patel R, Jain S, Aitken KL, Franks KN, van As N, Tree A, Hatfield P, Harrow S, McDonald F, Ahmed M, Saran FH, Webster GJ, Khoo V, Landau D, Eaton DJ, Hawkins MA. UK Consensus on Normal Tissue Dose Constraints for Stereotactic Radiotherapy. Clin Oncol (R Coll Radiol). 2018 Jan;30(1):5-14. doi: 10.1016/j.clon.2017.09.007. Epub 2017 Oct 13. PMID 29033164